CLINICAL TRIAL: NCT01931592
Title: Controling Intestinal Colonization of High Risk Patients With Extended Spectrum ß-Lactamase Producing Enterobacteriaceae (ESBL-E) - A Randomized Trial (CLEAR)
Brief Title: Controling Intestinal Colonization With Extended Spectrum ß-Lactamase Producing Enterobacteriaceae ESBL-E
Acronym: CLEAR
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: One of the study drugs was no longer available on a worldwide level.
Sponsor: Maria J.G.T. Vehreschild (Other)
Responsible Party: Sponsor-Investigator, Maria J.G.T. Vehreschild, Dr. med., University of Cologne
Organization: University of Cologne (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Uni-Koeln-1667
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Cancer
Keywords: ESBL; neutropenia; eradication; bloodstream infection; immunosuppression
MeSH Terms: conditions — Neoplasms; Neutropenia; Sepsis | interventions — Colistin; Gentamicins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ESBL eradication regimen (Active Comparator): Fosfomycin-trometamol (3 g granules dissolved in 200 ml of water for oral administration every 72h) and colistin (2x106 IU oral solution dissolved in 50-100 ml of water given orally every 6 hours) and gentamicin (an 80 mg oral solution dissolved in 50-100 ml of water given orally every 6 hours) will be administered in a double-blind fashion for a total duration of 7 days (day 1-7). The placebo treatment will be identical in taste, consistency, colour and packaging. To include the oral cavity into the eradication regimen, all medications should be gargled for at least 10 seconds before being swallowed.
  Interventions: Drug: ESBL eradication regimen
- Placebo ESBL eradication (Placebo Comparator): Placebo preparations of fosfomycin, gentamicin and colisitin, identical in taste, texture and color will be administered at the same rate as the active comparator medication.
  Interventions: Drug: Placebo ESBL eradication

INTERVENTIONS:
Drug: ESBL eradication regimen — Fosfomycin-trometamol (3 g granules dissolved in 200 ml of water for oral administration every 72h) and colistin (2x106 IU oral solution dissolved in 50-100 ml of water given orally every 6 hours) and gentamicin (an 80 mg oral solution dissolved in 50-100 ml of water given orally every 6 hours) will be administered in a double-blind fashion for a total duration of 7 days (day 1-7). The placebo treatment will be identical in taste, consistency, colour and packaging. To include the oral cavity into the eradication regimen, all medications should be gargled for at least 10 seconds before being swallowed.
  Other Names: fosfomycin-trometamol 3 g; colistin (2x106 IU; gentamicin (an 80 mg
  Arms: ESBL eradication regimen
Drug: Placebo ESBL eradication — Placebo preparations of fosfomycin, gentamicin and colisitin, identical in taste, texture and color will be administered at the same rate as the active comparator medication.
  Other Names: placebo preparations
  Arms: Placebo ESBL eradication

SUMMARY:
Rapid and rational health-care interventions are of great importance to efficiently combat the emergence of resistant and virulent bacteria. In recent years, spread of ESBL-E on a global level has been observed.

For ESBL-E, effective eradication regimens are not yet available. The current study therefore aims to assess a new approach to ESBL-E eradication. To avoid administration of the eradication regimen to patients at low risk of subsequent BSI with ESBL-E, the study population will be restricted to immunocompromised high-risk patients.

DETAILED DESCRIPTION:
Bloodstream infections (BSI) with multi-drug resistant (MDR) bacteria such as extended- spectrum betalactamase producing Enterobacteriaceae (ESBL-E) are associated with significant morbidity and mortality, particularly in the immunocompromised patient. In recent years, rapid spread of ESBL-E on a global level has been observed. While guidelines on effective infection control and treatment measures are urgently needed, the required basis of evidence is yet to be generated. Particularly data from interventional trials is lacking.

From October 2011 to December 2012, a multicenter cohort study on ESBL-E colonization and infection in haematology/oncology patients has been conducted within the Deutsches Zentrum für Infektionsforschung (DZIF) and allowed for a detailed description of the epidemiology of ESBL-E in this patient population. Based on these results, the sample size calculations for this study were carried out.

Rapid and rational health-care interventions are of great importance to efficiently combat the emergence of resistant and virulent bacteria. In recent years, spread of ESBL-E on a global level has been observed.

In 2012, the KRINKO (Kommission für Krankenhaushygiene und Infektionsprävention) at the Robert Koch Institute in Berlin, German, published their new recommendations on the management of colonization and infection with Gram-negative MDR bacteria, including ESBL-E. In high-risk settings, e.g. haematology/oncology wards and intensive care units, contact isolation is recommended for all patients who are colonized or infected with ESBL-E. While recommendations of the KRINKO are not legally binding, many institutions are now integrating these suggestions into their standards of care, given the recent increase in the prevalence of ESBL-E. This development is putting a considerable strain on patients and treating physicians. Firstly, previous studies have demonstrated the negative impact of long-term isolation on the patients' frequency of contacts with health care workers, a decrease in scores for self-esteem and an increase in scores for anxiety and depression.Secondly, proper contact isolation requires treatment in a single room. Many hospitals are, however, not equipped with sufficient numbers of single rooms, to accommodate all patients carrying MDR bacteria. Apart from problems associated with contact isolation, immunocompromised patients who are colonized with ESBL-E are at an increased risk of subsequent bloodstream infections (BSI).

Medical care providers are used to be faced with similar problems when dealing with methicillin-resistant Staphylococcus aureus (MRSA). However, nowadays, eradication regimens offer the possibility to remove MRSA from the skin and mucosa of colonized patients, thus interrupting its further spread to a considerable extent. For ESBL-E, effective eradication regimens are not yet available. The current study therefore aims to assess a new approach to ESBL-E eradication. To avoid administration of the eradication regimen to patients at low risk of subsequent BSI with ESBL-E, the study population will be restricted to immunocompromised high-risk patients.

The human intestinal tract is known to be colonized by hundreds of different bacterial species and other microbes. Based on the experience with fecal microbiota therapy in the treatment of recurrent Clostridium difficile infections, it can be hypothesized that the intestinal microbiome may influence the success or failure of the present study intervention. Thus, at selected sites, a metagenomic analysis of the intestinal microbiome will be performed to explore possible associations between certain microbiome patterns and the successful eradication of ESBL-E.

There is an ongoing discussion on whether antibiotic regimens used for eradication and selective digestive tract decontamination (SDD) might lead to the emergence of multi-drug resistant bacteria.11 Emergence of resistance under long-term administration of SDD to ICU patients has been previously reported.12 However, a recently published meta-analysis, including 64 studies in ICUs, of which 47 were randomized controlled trials and 35 included data for the detection of antimicrobial resistance, no relation between the use of SDD and the development of antimicrobial resistance could be detected.13 Even without this information, the risk for emergence of resistance should be classified as very low, considering that patients will receive eradication treatment for the duration of only seven days. Nevertheless, the possible emergence of non-ESBL multi-drug resistant bacteria in the intestine will be assessed during the study intervention.

Concerning the choice of an antibiotic regimen with a high chance of effectively eradicating ESBL-E from the gut, data from previous studies has been taken into account. Most previous study concepts were based on the idea of SDD.14-16 SDD aims to eradicate abnormal aerobic gram-negative bacteria, while preserving anaerobic bacteria. In this setting, the problem of adverse events caused by systemic effects of the antibiotics used can be discarded. However, if only locally active antibiotics are used for achieving eradication, patients are less likely to clear concurrent ESBL-E colonization of the throat, skin and urinary bladder. These body sites may then serve as a source of intestinal re-colonization with ESBL-E. Therefore, the current pilot study uses a combination of a non-absorbable enterally administered antibiotic and a systemic antibiotic. To facilitate the choice of an optimum non-absorbable antibiotic, antimicrobial susceptibility testing of clinical isolates of ESBL-E from haematological high-risk patients was carried out at the University Hospital Cologne in 2012. Virtually no resistance towards colistin could be detected (data not published), such that colistin was chosen as the non-absorbable component. As previous studies have shown promising results for a combination of colistin and gentamicin, the latter was added to the eradication regimen. Concerning the choice of a systemically active antibiotic, promising data on the clinical efficacy of fosfomycin in ESBL-E infections and in the reduction of ESBL-E in the intestinal flora have been published. Given the additional convenience of an available oral formulation - a prerequisite not given for most other ESBL-E active treatments - fosfomycin was chosen for combination with oral colistin and gentamicin. For the treatment of urinary tract infections, oral fosfomycin is usually administered as a single dose of 3g. However, several studies have assessed treatment of complicated or chronic urinary tract infections with repetitive administrations of 3g fosfomycin.

Since a single dose may not suffice to reduce the intestinal ESBL-E burden below the limit of detection, a schedule of 3g p.o. every 72h was chosen for this study.

ELIGIBILITY:
Inclusion Criteria:

* Fecal colonization with ESBL-E, as confirmed by a positive sample (rectal swab or stool sample) obtained within 14 days prior to study enrolment
* Ongoing or scheduled immunosuppression:

  * allogeneic or autologous hematopoietic stem cell transplantation within 14 days after enrollment or
  * chemotherapy with an expected duration of chemotherapy-associated neutropenia of at least 7 days within 14 days after enrollment or
  * solid organ transplantation within 14 days after enrollment or
  * administration of high-dose corticosteroids or other immunosuppressants for acute rejection of a solid organ transplant or for graft versus host disease after stem cell transplantation
* Age of at least 18 years
* Subject is not legally incapacitated
* Written informed consent from the trial subject has been obtained

Exclusion Criteria:

* Current or scheduled administration of ESBL-E active antibiotic treatment after receipt of the most recent sample showing intestinal ESBL-E colonization and within 10 days after randomization
* Planned selective digestive tract decolonization within 42 days following randomization
* Known hypersensitivity or allergy to any of the components of the study treatment
* Moderate or severe liver dysfunction at baseline, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels greater than three times the upper limit of normal (ULN), AND a total bilirubin level greater than two times the ULN
* Serum creatinine > 2 x the upper limit of the ULN
* Inability to take oral medication
* Concurrent participation in another clinical trial with an investigational drug is not permitted, unless the drug under study is related to the treatment of the underlying condition or a transplantation
* Current pregnancy or nursing period
* In female study participants, failure to use highly-effective contraceptive methods. The following contraceptive methods with a Pearl Index lower than 1% are regarded as highly-effective:

  * Oral hormonal contraception ('pill')
  * Dermal hormonal contraception
  * Vaginal hormonal contraception (NuvaRing®)
  * Contraceptive plaster
  * Long-acting injectable contraceptives
  * Implants that release progesterone (Implanon®)
  * Tubal ligation (female sterilization)
  * Intrauterine devices that release hormones (hormone spiral)
  * Double barrier methods This means that the following are not regarded as safe: condom plus spermicide, simple barrier methods (vaginal pessaries, condom, female condoms), copper spirals, the rhythm method, basal temperature method, and the withdrawal method (coitus interruptus).
* Patient has any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of the patient participating in the study, would make it unlikely for the patient to complete the study, or would confound the results of the study
* Persons with any kind of dependency on the investigator or employed by the sponsor or investigator
* Persons held in an institution by legal or official order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-01; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Short-term intestinal eradication | 11 days
  Short-term intestinal eradication, defined as a fecal sample , negative for ESBL-E on day 6+/-1 and day 11+/-2

SECONDARY OUTCOMES:
Long-term intestinal eradication d28 | 28 days
  Long-term intestinal eradication d28, defined as a fecal sample1, negative for ESBL-E on day 28+/-4
Long-term intestinal eradication d42 | 42 days
  Long-term intestinal eradication d42, defined as a fecal sample1, negative for ESBL-E on day 42+/-4
Short-term non-intestinal eradication | 11 days
  Short-term non-intestinal eradication, defined as a combination of ESBL-E negative samples from urine and throat on day 6+/-1 and day 11+/-2
Long-term non-intestinal eradication d28 | 28 days
  Long-term non-intestinal eradication d28, defined as a combination of ESBL-E negative samples from urine and throat on day 28+/-4
Long-term non-intestinal eradication d42 | 42 days
  Long-term non-intestinal eradication d42, defined as a combination of ESBL-E negative samples from urine and throat on day 42+/-4
Emerging presence of non-ESBL multi-drug resistant bacteria | 42 days
  Emerging presence of non-ESBL multi-drug resistant bacteria in the intestine, defined as identification of vancomycin resistant Enterococci (VRE), carbapenem- resistant gram negative rods (4MRGN according to the KRINKO definition) or colistin-resistant enterobacteria (except Proteus and Serratia spp.) in a fecal sample on day 6+/-1, day 11+/-2, day 28+/-4 or day 42+/-4
Intestinal microbiome | 42 days
  Association between the intestinal microbiome pattern and the outcome of eradication on baseline, day 6+/-1, day 11+/-2, day 28+/-4 or day 42+/-4
Quantitative assessment of intestinal ESBL-E burden | 42 days
  Quantitative assessment of intestinal ESBL-E burden on baseline, day 6+/-1, day 11+/-2, day 28+/-4 or day 42+/-4
Incidence and severity of AEs | 42 days
  Incidence and severity of AEs
Rate of AE-related study drug discontinuations | 42 days
  Rate of AE-related study drug discontinuations

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Vehreschild, MD, Principal Investigator — University Hospital Cologne
Locations (2):
- Germany (2):
  - University hospital Hamburg Eppendorf, Hamburg, Hamburg
  - University Hospital Cologne, Cologne, North Rhine-Westphalia

REFERENCES:
- [Derived] Dimitriou V, Biehl LM, Hamprecht A, Vogel W, Dorfel D, Peter S, Schafhausen P, Rohde H, von Lilienfeld-Toal M, Klassert TE, Slickers P, Ehricht R, Slevogt H, Christ H, Hellmich M, Farowski F, Tsakmaklis A, Higgins PG, Seifert H, Vehreschild MJGT. Controlling intestinal colonization of high-risk haematology patients with ESBL-producing Enterobacteriaceae: a randomized, placebo-controlled, multicentre, Phase II trial (CLEAR). J Antimicrob Chemother. 2019 Jul 1;74(7):2065-2074. doi: 10.1093/jac/dkz124. PMID 31220256